CLINICAL TRIAL: NCT03339518
Title: BRIM3: Breast Cancer Recurrence Risk Informational Materials Project
Brief Title: Breast Cancer Recurrence Risk Counseling
Acronym: BRIM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Kimberly Kelly, Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1306056017
Record Dates: First submitted 2017-10-24; First posted 2017-11-13 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIM3 Educational intervention (Experimental): Individuals will receive a booklet and counseling about risk.
  Interventions: Behavioral: BRIM3 educational intervention
- Wait list Control (Other): At the completion of the study, individuals in the wait list condition will receive a booklet.
  Interventions: Behavioral: Wait List

INTERVENTIONS:
Behavioral: BRIM3 educational intervention — Breast Cancer risk education and counseling
  Arms: BRIM3 Educational intervention
Behavioral: Wait List — Booklet at the end of study
  Arms: Wait list Control

SUMMARY:
The number of breast cancer survivors is growing. Women with a personal history of breast cancer worry about their risk of getting cancer again. The current study will develop counseling about breast cancer recurrence risk and will also get an estimate of the preliminary impact of this counseling. The goal is to enable women to make better decisions about their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women who (1) have a personal history of a single stage 0-2 breast cancer, (2) were recently diagnosed within the past 6 months, and (3) are treated at a participating breast oncology clinic.

Exclusion Criteria:

* Women who are unable to read/write in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2011-07-25 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Comparative Perceived Risk of Breast Cancer | 6 months
  Comparative perceived risk will be assessed with a comparative risk item (i.e., compared those of the same gender and race; Lipkus, CEBP 2000).
Absolute Perceived Risk of Breast Cancer | 6 months
  Absolute perceived risk will be assessed with an absolute risk item to assess risk as a percentage (Kelly, PONC, 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kelly, PhD, Principal Investigator — 304-293-1453
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be available upon written request is appropriate human subjects protections are in place, and the request does not conflict with the aims of the study.